CLINICAL TRIAL: NCT03146286
Title: Skeletal Muscle Protein Metabolism and Insulin Sensitivity in Overweight Individuals: Effects of Meals With Various Fatty Acid Compositions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SCA/OF/12/15
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Fatty Acids; Fish Oils

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Chocolate flavoured drink spiked with 15mg/kg [2H31]palmitate (D31palmitate) and singly-labelled water (H218O). 4 hours post test meal a bolus of milk protein (30 g), which has been intrinsically labelled with [13C]phenylalanine, along with 75 g of glucose in 250 ml of water will be given.
  Interventions: Dietary Supplement: Placebo
- Saturated Fat (Experimental): Chocolate flavoured drink spiked with 15mg/kg [2H31]palmitate (D31palmitate) and singly-labelled water (H218O) containing 0.7 g/kg bodyweight palm stearin. 4 hours post test meal a bolus of milk protein (30 g), which has been intrinsically labelled with [13C]phenylalanine, along with 75 g of glucose in 250 ml of water will be given.
  Interventions: Dietary Supplement: Saturated fat
- Fish Oil (Experimental): Chocolate flavoured drink spiked with 15mg/kg [2H31]palmitate (D31palmitate) and singly-labelled water (H218O) containing 0.45 g/kg bodyweight palm stearin and 0.25 g/kg bodyweight fish oil (n3PUFA). 4 hours post test meal a bolus of milk protein (30 g), which has been intrinsically labelled with [13C]phenylalanine, along with 75 g of glucose in 250 ml of water will be given.
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Saturated fat — Palm stearin
  Arms: Saturated Fat
Dietary Supplement: Placebo — Water
  Arms: Control
Dietary Supplement: Fish Oil — Fish Oil, Omega 3 PUFA
  Arms: Fish Oil

SUMMARY:
The aim of the study will investigate whether impairment in the action of insulin to promote the use of glucose in skeletal muscle (insulin resistance) as a result of oral ingestion of a liquid meal rich in saturated fat is linked to reduced ability of muscles to synthesise new protein in response to dietary protein intake, which ultimately may compromise maintenance of muscle size and quality of life and whether partially replacing saturated fat in the liquid meal with omega 3 polyunsaturated FA (n3PUFA) will ameliorate these negative effects.

ELIGIBILITY:
Inclusion Criteria:

* Male, healthy, overweight (BMI>27 kg/m2 and fat mass >30%) non-diabetic individuals.

Exclusion Criteria:

* Diabetes, smoking, cardiovascular disease

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2015-12-03 (Actual); Study Completion 2015-12-03 (Actual)

PRIMARY OUTCOMES:
Change in muscle protein fractional synthetic rate | 3 hours post protein drink
  Measurement of FSR at baseline and post intervention

SECONDARY OUTCOMES:
whole body postprandial insulin sensitivity | Baseline and every 15mins for 7 hours
  Glucose and insulin area under the curves (AUC) in response to the milk protein and glucose ingestion will be measured
Whole body and skeletal muscle fat oxidation | Baseline and every 15mins for 7 hours
  D31palmitate plasma enrichment and incorporation into skeletal muscle lipids

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jans A, Konings E, Goossens GH, Bouwman FG, Moors CC, Boekschoten MV, Afman LA, Muller M, Mariman EC, Blaak EE. PUFAs acutely affect triacylglycerol-derived skeletal muscle fatty acid uptake and increase postprandial insulin sensitivity. Am J Clin Nutr. 2012 Apr;95(4):825-36. doi: 10.3945/ajcn.111.028787. Epub 2012 Feb 15. PMID 22338035
- [Background] Newens KJ, Thompson AK, Jackson KG, Wright J, Williams CM. DHA-rich fish oil reverses the detrimental effects of saturated fatty acids on postprandial vascular reactivity. Am J Clin Nutr. 2011 Sep;94(3):742-8. doi: 10.3945/ajcn.110.009233. Epub 2011 Aug 10. PMID 21831993
- [Background] Nowotny B, Zahiragic L, Krog D, Nowotny PJ, Herder C, Carstensen M, Yoshimura T, Szendroedi J, Phielix E, Schadewaldt P, Schloot NC, Shulman GI, Roden M. Mechanisms underlying the onset of oral lipid-induced skeletal muscle insulin resistance in humans. Diabetes. 2013 Jul;62(7):2240-8. doi: 10.2337/db12-1179. Epub 2013 Mar 1. PMID 23454694
- [Derived] Wilhelmsen A, Davies A, Mallinson J, Pabla P, Jones R, Palmer EA, Dunn WB, Moran GW, Stephens FB, Tsintzas K. Acute effects of prior dietary fat ingestion on postprandial metabolic responses to protein and carbohydrate co-ingestion in overweight and obese men: A randomised crossover trial. Clin Nutr. 2022 Aug;41(8):1623-1635. doi: 10.1016/j.clnu.2022.06.022. Epub 2022 Jun 16. PMID 35764009